CLINICAL TRIAL: NCT05415085
Title: Culprit-first Versus Culprit-last Approach During Primary Percutaneous Coronary Intervention in Patients With ST-elevation Myocardial Infarction: A Randomized Controlled Study
Brief Title: Culprit-first in Primary Percutaneous Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Nir Levi, Physician, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2022-04-27; First posted 2022-06-10 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease; Myocardial Infarction; STEMI; Stent
Keywords: coronary artery disease; STEMI; primary PCI; door-to-balloon time
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culprit-first PCI (Experimental): In this arm, primary PCI with stent implantation will be performed prior to the demonstration of the whole coronary tree. The suspected culprit artery will be demonstrated first and the PCI will be performed.
  Interventions: Procedure: Culprit-first PCI
- Culprit-last PCI (No Intervention): In this arm, primary PCI with stent implantation will be performed after the demonstration of the whole coronary tree. The suspected culprit artery will be demonstrated after the contralateral side and then PCI will be performed. This is the common approach.

INTERVENTIONS:
Procedure: Culprit-first PCI — PCI to the culprit artery prior to the demonstration of the whole coronary tree.
  Arms: Culprit-first PCI

SUMMARY:
The aim of this study is to assess the impact of culprit-first versus culprit-last percutaneous coronary intervention on the door to balloon time and clinical outcomes in patients with ST-elevation myocardial infarction.

DETAILED DESCRIPTION:
Ischemic heart disease (IHD) is the single most common cause of death and its frequency is increasing globally. It is estimated that IHD is the cause of 1.8 million deaths or 20% of all deaths in Europe. Despite advancements in the fields of rapid diagnosis and in treatment strategies, the morbidity, and mortality in patients with ST-segment myocardial infarction remains substantial, with an estimated mortality rate of 4-12% according to registries of the ESC countries. According to the 2017 European Society of Cardiology (ESC) guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation (STEMI), there is a level 1 recommendation with a level of evidence A for primary percutaneous coronary intervention (PPCI) strategy in patients with STEMI, and this strategy is preferred over fibrinolytic therapy. In addition, the ESC guidelines recommend a first medical contact to reperfusion time within 60 minutes in STEMI patients for primary PCI-capable centers. This recommendation is supported by a recently published study that showed shortening door to balloon (D2B) time was significantly associated with survival benefit. Based on the recommendation for maximal D2B time in STEMI patients to be 60 minutes, many countries and institutions worldwide have established programs, among them the national program for quality indicators by the Israeli ministry of health, to shorten D2B times. According to data published by the Israeli ministry of health in the year 2018, 88% of STEMI patients had a D2B time of <90 minutes. The common practice during PPCI is to complete diagnostic angiography of the whole coronary tree before performing culprit-vessel revascularization. This practice is not evidence-based and current guidelines do not prioritize full diagnostic angiography over culprit-vessel revascularization first. As was found in previous studies, this practice might result in delaying revascularization by 4-8 minutes in D2B time. This delay might potentially lead to worse outcomes in STEMI patients, although not proven in the above-cited studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with STEMI who are eligible for PPCI

Exclusion Criteria:

* Cardiac arrest
* Cardiopulmonary resuscitation or extracorporeal membrane oxygenation on arrival to the catheterization laboratory
* Prior coronary artery bypass grafting surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Needle-to-balloon time of 10 minutes or less | through study completion, an average of 1 year
  Change in needle-to-balloon time in minutes

SECONDARY OUTCOMES:
Need for hemodynamic (mechanical/medical) support during PCI | through study completion, an average of 1 year
  Number of patients that needed mechanical support during PCI
Need for respiratory support during PCI | through study completion, an average of 1 year
  Number of patients that needed respiratory support during PCI
Rate of failed PCI | through study completion, an average of 1 year
  As determined by the operator

CONTACTS AND LOCATIONS:
Overall Officials: Nir Levi, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levi N, Wolff R, Jubeh R, Shuvy M, Steinmetz Y, Perel N, Maller T, Amsalem I, Hitter R, Asher E, Turyan A, Karmi M, Orlev A, Dratva D, Khoury Z, Hasin T, Wolak A, Glikson M, Dvir D. Culprit Lesion Coronary Intervention Before Complete Angiography in ST-Elevation Myocardial Infarction: A Randomized Clinical Trial. JAMA Netw Open. 2024 Mar 4;7(3):e243729. doi: 10.1001/jamanetworkopen.2024.3729. PMID 38551563